CLINICAL TRIAL: NCT03437122
Title: Project A3sc - An Atlas of Airways at a Single Cell Level
Acronym: AAAsc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-PP-14
Record Dates: First submitted 2018-01-17; First posted 2018-02-19 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Respiratory System
Keywords: lung, nasal mucosa, respiratory mucosa
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All (Experimental)
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Multiple level sampling of the respiratory mucosa (cytology brush and biopsies forceps)

SUMMARY:
The increasing incidence of chronic respiratory diseases is a public health problem affecting hundreds of thousands of people around the world, including children. Directly exposed to atmospheric aerocontaminants (pollution, allergens), the respiratory tracts represent a complex ecosystem that involves different cells that develop complex interactions with the surrounding connective tissue but also with their rich immune environment and with the microbiota. Although a pathophysiological continuum is postulated between the nasal and bronchial airways in certain diseases, such as allergic diseases, we have identified broad gradients in gene expression between nasal and bronchial samples. This is why cellular variability throughout the respiratory tree needs to be studied in detail.

The sequencing of RNAs specifically present in a particular cell, and its comparison with neighboring cells, allows us to document precise cellular contributions and intercellular relationships. Our project will establish protocols to stabilize airway swabs by brushing and/or biopsy, under conditions that will then allow the analysis of gene expression profiles at the single cell level (single cell RNA sequencing).

The development of the "single cell" stabilisation and analysis protocol will first be carried out on primary respiratory epithelium cultures and then extended to respiratory specimens taken from healthy volunteers. Through sampling at several levels of the respiratory tree, variations in expression along the tracheobronchial axis will be fully documented. Finally, the interaction between the epithelial compartment and the immunological compartment will be studied by analyzing gene expression on a single cell in different physiopathological contexts.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years and <40 years
* non-smoker
* absence of known acute or chronic disease
* absence of symptoms suggestive of progressive disease
* normal clinical examination

Exclusion Criteria:

* recent rhino-bronchial infection (<6 weeks)
* mental disability
* pregnant women (a urine test will be performed for all women of childbearing age)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Number of samples usable | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie LEROY, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No